CLINICAL TRIAL: NCT00507546
Title: Melatonin Replacement for Treatment of Sleep Disruption
Brief Title: Functional Melatonin Replacement for Sleep Disruptions in Individuals With Tetraplegia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Stanford University (Other); Takeda (Industry)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B6010-R; 06-038R (Other Grant/Funding Number: VA)
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Results first posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-04

CONDITIONS: Insomnia; Spinal Cord Injury; Tetraplegia; Sleep Disorders
Keywords: sleep; melatonin; spinal cord injury; insomnia; tetraplegia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Spinal Cord Injuries; Quadriplegia; Sleep Wake Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon then placebo (Experimental): 8 mg nightly ramelteon for three weeks, followed by two weeks of nightly placebo (washout), then three weeks of nightly placebo (cross-over)
  Interventions: Drug: Ramelteon
- Placebo then ramelteon (Experimental): placebo nightly for three weeks, followed by two weeks of nightly placebo (washout), then three weeks of 8 mg nightly ramelteon (cross-over)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — 8 mg nightly
  Other Names: Rozerem
  Arms: Ramelteon then placebo
Drug: Placebo — Nightly 8mg of placebo (same appearance as ramelteon)
  Arms: Placebo then ramelteon

SUMMARY:
The purpose of this study is to determine if replacing melatonin function with a melatonin agonist (ramelteon) in individuals that lack endogenous melatonin production (tetraplegia) helps to alleviate self-reported sleep disruption.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older, male or female veterans of any racial or ethnic group
* Neurologically complete (Frankel A or B) damage to the lower (C4-C8) cervical spinal cord
* Absence of melatonin production
* Time since SCI is greater than 6 months [no cases of acute spinal cord injury]
* Subjective complaint of sleep disruption

Exclusion Criteria:

* Current use of fluvoxamine (Luvox , antidepressant), rifampin (antimycobacterial), ketoconazole (Nizoral , antifungal), or fluconazole (Diflucan , antifungal) [these interact with the same liver enzyme that is the primary metabolizer of ramelteon]; use of sleep medications is okay
* Hepatic dysfunction
* Concomitant use of over-the-counter melatonin
* Pregnancy or breast feeding
* Currently or have within the past six months met DSM-IV (Diagnosis and Statistical Manual IV) criteria for drug or alcohol abuse or dependence or AUDIT score >19
* Acute illness or unstable chronic illness. Use of continuous positive airway pressure (CPAP) for treatment of sleep apnea is acceptable.
* No travel across three or more time zones within three weeks or during the protocol
* Illiterate or unable to read or write English or are judged by the investigator to be unable or unlikely to follow the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M. Zeitzer, PhD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Result] Zeitzer JM, Ku B, Ota D, Kiratli BJ. Randomized controlled trial of pharmacological replacement of melatonin for sleep disruption in individuals with tetraplegia. J Spinal Cord Med. 2014 Jan;37(1):46-53. doi: 10.1179/2045772313Y.0000000099. Epub 2013 Oct 24. PMID 24090266

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from community
Pre-assignment Details: Subjects excluded if baseline measure detected the presence of melatonin metabolite in their urine.
Groups:
- Arm 1: Ramelteon then placebo
  Ramelteon : 8 mg nightly
- Arm 2: Placebo then ramelteon
  Placebo : Nightly 8mg of placebo (same appearance as ramelteon)
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 4 | 4
Completed | 2 | 3
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.25 (9.74) | 55.5 (15.5) | 53 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Amount of Wakefulness After Sleep Onset (WASO)
Description: Measured as the median of the average WASO of the three weeks of either placebo or ramelteon treatment
Time Frame: 10 weeks
Population: All participants who completed the entire protocol.
Measure: Median (Full Range); unit: Minutes
Groups:
- Ramelteon: Ramelteon then placebo
  Ramelteon : 8 mg nightly
- Placebo: Placebo then ramelteon
  Placebo : Nightly 8mg of placebo (same appearance as ramelteon)
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 3 | 2
Minutes | 72.3 [20.7 to 92.3] | 76.5 [24.0 to 117]
Statistical Analysis 1: Comparison: Ramelteon vs Placebo; Test type: Superiority or Other; p = 0.70, Friedman

2. Secondary Outcome: Change in Subjective Morning Alertness
Description: Measured as the median of the average morning alertness (measured from 1-7 on the Stanford Sleepiness Scale, a Likert-like scale in which higher values are lower alertness) of the three weeks of either placebo or ramelteon treatment
Time Frame: 10 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 3 | 2
units on a scale | 2.86 [2.05 to 3.57] | 3.14 [1.15 to 5.83]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = 0.35, Friedman

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No